CLINICAL TRIAL: NCT06823895
Title: Exploring the Pharmacokinetics of Oligonucleotides in Maixuekang Capsules in Healthy Subjects
Brief Title: Pharmacokinetic Study of Oligonucleotides in Maixuekang Capsules
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NFEC-2024-383
Record Dates: First submitted 2024-12-15; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-dose (Experimental): Maixuekang capsules, once, 1g, orally
  Interventions: Drug: Maixuekang capsule
- multiple-dose (Experimental): Maixuekang capsules，1g each time, 3 times/day, 3 days, orally
  Interventions: Drug: Maixuekang capsule

INTERVENTIONS:
Drug: Maixuekang capsule — Single dose group: Participants will be given Maixuekang capsules once, 1g, orally.
  Multiple dose group: Participants will receive 1g of Maixuekang capsules orally for 3 days, 3 times a day.

SUMMARY:
The objective of this clinical trial is to learn the sequence and expression level of Maixuekang oligonucleotides in the plasma of healthy volunteers.

1. Detecting the sequence and expression levels of oligonucleotides in the blood of healthy subjects before and after a single administration of Maixuekang at different time points.
2. Detecting the sequence and expression levels of oligonucleotides in the blood of healthy subjects before and after multiple administrations of Maixuekang at different time points.

Single dose group: Participants will be given Maixuekang capsules once, 1g, orally.

Multiple dose group: Participants will receive 1g of Maixuekang capsules orally for 3 days, 3 times a day.

DETAILED DESCRIPTION:
This study is an exploratory study of the active substances in the marketed drug "Maixuekang Capsule". "Maixuekang Capsule" is a traditional Chinese patent medicines and simple preparations approved by the State Food and Drug Administration of China, which has been used for more than 20 years. It is made of live leeches through freeze-dried, containing protein and nucleotide of animal tissues.

In this study, the investigators will explore the sequence and expression levels of oligonucleotides in the plasma of healthy subjects in Maixuekang capsules at different time points before and after single and multiple administrations.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy subjects aged 18 to 45 years (including the critical value);
2. Male weight ≥ 50.0kg, female weight ≥ 45.0kg; Body mass index (BMI) ranges from 19.0 to 26.0 kg/m2 (including boundary values);
3. Normal or abnormal medical history, vital signs, physical examination, clinical laboratory tests (including blood routine, urine routine, blood biochemistry, coagulation function test), 12 lead electrocardiogram, etc. have no clinical significance;
4. The subjects and their partners were able to take effective contraceptive measures during the trial period and did not have any fertility plans during the trial period or within 6 months after the trial ended;
5. The subjects fully understand the content, process, and possible adverse reactions of the experiment and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Any previous cause or disease that leads to thrombocytopenia, coagulation dysfunction, or bleeding tendency, including recurrent gum bleeding, peptic ulcers, severe or long-term heavy menstrual flow, etc;
2. Those who are allergic to heterologous animal proteins and leeches;
3. Individuals who have a smoking habit within the previous 3 months (averaging over 5 cigarettes per day) or who cannot stop using any tobacco products throughout the entire trial period after being selected;
4. Screening for those who have been addicted to alcohol within the past 3 months (drinking more than 14 units of alcohol per week: 1 unit=285mL of beer, 25mL of spirits, or 100mL of wine) or have consumed any alcoholic products or alcohol breath tests positive within 24 hours before administration, or those who cannot accept the prohibition of drinking throughout the entire trial period after being selected;
5. Those who have consumed excessive amounts of tea, coffee, or beverages containing caffeine within the past 3 months, or have consumed any food or beverage containing caffeine (such as coffee, strong tea, chocolate, etc.) or xanthine (such as dragon fruit, mango, etc.) or citrus fruits of the Rutaceae family (such as grapefruit, etc.) within 48 hours before administration;
6. Those who have participated in drug trials and taken the investigational drug within 3 months prior to the screening period, or those who have participated in medical device research within 3 months of the screening period;
7. Patients who have difficulty swallowing or have any diseases (whether cured or not) or surgeries (excluding appendectomy) that affect drug absorption, distribution, metabolism, and excretion, as well as gastric motility and pH value, within the 6 months prior to screening, or who plan to undergo surgery during the study period;
8. Have a history of drug abuse or tested positive for drug abuse within the past 6 months prior to screening;
9. Individuals who have tested positive for drug screening or have a history of drug abuse within 5 years prior to their first use of the study drug, or have used drugs within 3 months prior to their first use of the study drug;
10. Individuals who are positive for hepatitis B surface antigen, Treponema pallidum antibody, human immunodeficiency virus antibody, and hepatitis C antibody;
11. Pregnant and lactating women or those whose blood β - HCG test is positive;
12. Acute illness or concomitant medication occurs from the screening stage to the study medication;
13. Difficulty in venous blood collection, or inability to tolerate venipuncture blood collection, or a history of dizziness or needle fainting;
14. Those who cannot follow a uniform diet (such as having special dietary requirements, intolerance to standard meal foods, etc.);
15. The researcher determines that the subjects have any other circumstances that make them unsuitable to participate in this clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perform UMI Small RNA sequencing on blood samples at different time points | Single dose group: within 1 hour before administration, 3 hours, 3.5 hours, 4 hours, 6 hours, 8 hours, and 12 hours after administration; Multiple dose group: within 1 hour before the first administration, 10 hours, 16 hours, 28 hours, 40 hours
  "Maixuekang Capsule" is a traditional Chinese patent medicines and simple preparations approved by the State Drug Administration of China, which has been used for more than 20 years. It is made of leeches through freeze drying.
  This project will collect blood samples before administration, as well as at 3, 3.5, 4, 6, 8, and 12 hours after administration. Unique Molecular Identifier small RNA Seq sequencing technology will be used to detect the small RNA sequences of the blood samples and compare them with the leech genome to identify which leech specific small RNA sequences have entered human blood, as well as the table of these sequences at different time points after administration

SECONDARY OUTCOMES:
Adverse event rate | Single dose group: within 24 hours of administration; Multi dose group: within 5 days after the first administration.
  Number of participants with With Treatment-Related Adverse Events as Assessed by CTCAE v5.0, with abnormal vital signs, abnormal physical examination, abnormal 12 lead electrocardiogram, and abnormal laboratory tests results

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, China